CLINICAL TRIAL: NCT05973305
Title: A Randomized, Open-label, Controlled, Comparative Study of Efficacy and Safety of Dorzol Eye Drops, 20 mg/mL (JGL dd, Croatia) vs Trusopt® Eye Drops, 20 mg/mL (Merck Sharp & Dohme, France) in Patients With Primary Open-angle Glaucoma
Brief Title: Comparative Study of Dorzol Eye Drops, 20 mg/ml Versus Trusopt® Eye Drops, 20 mg/ml
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Jadran Galenski laboratorij d.d. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DORZOL-10/2015
Record Dates: First submitted 2023-07-26; First posted 2023-08-02 (Actual); Last update posted 2023-08-02 (Actual); Status verified 2023-04

CONDITIONS: Primary Open Angle Glaucoma of Both Eyes
Keywords: Glaucoma; Intraocular pressure; Treatment
MeSH Terms: conditions — Glaucoma | interventions — dorzolamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patients with primary open-angle glaucoma receiving Dorzol 20 mg/ml (Experimental): Dorzol 20 mg/ml eye drops, dosing schedule t.i.d, 12 weeks
  Interventions: Drug: Dorzol 20 mg/ml
- Patients with primary open-angle glaucoma receiving Trusopt 20 mg/ml (Active Comparator): Trusopt 20 mg/ml eye drops, dosing schedule t.i.d, 12 weeks
  Interventions: Drug: Trusopt 20 mg/ml

INTERVENTIONS:
Drug: Dorzol 20 mg/ml — dosing schedule t.i.d.
  Other Names: Dorzol
  Arms: Patients with primary open-angle glaucoma receiving Dorzol 20 mg/ml
Drug: Trusopt 20 mg/ml — dosing schedule t.i.d.
  Other Names: Trusopt
  Arms: Patients with primary open-angle glaucoma receiving Trusopt 20 mg/ml

SUMMARY:
The goal of this study is to compare efficacy and safety of Dorzol 20 mg/mL Eye Drops manufactured by JADRAN-GALENSKI LABORATORIJ d.d. (Croatia) aimed at lowering elevated IOP in patients with ocular hypertension and primary open-angle glaucoma (POAG) versus TRUSOPT 20 MG/ML Eye Drops manufactured by Laboratoires Merck Sharp & Dohme-Chibret, France. The main questions it aims to answer are:

* if the efficacy of the investigational drug and the reference drug in patients with ocular hypertension and primary open-angle glaucoma is equal;
* if the safety of the investigational drug and the reference drug in patients with ocular hypertension and primary open-angle glaucoma is equal.

A total of 118 participants were screened and randomized 1:1 to the investigational drug (Dorzol) group or the reference drug (Trusopt) group. 59 patients were recruited in each group.

Researchers compared the investigational drug (Dorzol) group with the reference drug (Trusopt) group to see if the efficacy and safety of the investigational drug and the reference drug in patients with ocular hypertension and primary open-angle glaucoma are equal.

DETAILED DESCRIPTION:
Study Title:

A randomized, open-label, controlled, comparative study of efficacy and safety of Dorzol eye drops, 20 mg/mL, manufacturer: JADRAN - GALENSKI LABORATORIJ d.d., Croatia, vs. Trusopt® eye drops, 20 mg/mL, manufacturer: Laboratoires Merck Sharp & Dohme-Chibret, France, in patients with primary open-angle glaucoma.

Protocol No. DORZOL-10/2015, version No. 1.0 of 25.10.2015 RCT No. 629 of 07.09.2016 Investigators

1. Abdulaeva Elmira Abdulaevna (Test facility No.4)
2. Eryomina Alyona Victorovna (Test facility No.6)
3. Lisitsyn Alexey Borisovich (Test facility No.7)
4. Doga Alexander Victorovich (Test facility No.8) Test facilities No.4. State autonomous healthcare institution 'Republican Clinical Ophthalmological Hospital of the Ministry of Health of the Republic of Tatarstan', 420012, Republic of Tatarstan, Kazan, Butlerova St., 14.

   No.6. Federal state autonomous institution 'Acad. S.N. Fyodorov Eye Microsurgery Interbranch Science and Technology Complex', Ministry of Health of the Russian Federation, 127486, Moscow, Beskudnikovsky Blvd., 59A.

   No.7. State healthcare institution of Yaroslavl region 'Clinical Hospital No. 8', 150030. Yaroslavl, Suzdalskoe Highway, 39.

   No.8. Federal state autonomous institution 'Acad. S.N. Fyodorov Eye Microsurgery Interbranch Science and Technology Complex', Ministry of Health of the Russian Federation, 127486, Moscow, Beskudnikovsky Blvd., 59A.

   Study period:

   First patient enrollment date: 5 April 2017 Study completion date: 1 September 2018 Phase III (a safety and efficacy study)

   Study objective:

   The study objective was to evaluate the efficacy and safety of Dorzol eye drops, 20 mg/mL, manufacturer: JADRAN - GALENSKI LABORATORIJ d.d., Croatia, designed to reduce elevated intraocular pressure in patients with primary open-angle glaucoma (POAG), vs. Trusopt® eye drops, 20 mg/mL, manufacturer: Laboratoires Merck Sharp & Dohme-Chibret, France.

   Study tasks:
   * Prove noninferiority of the test vs. reference product in patients with primary open-angle glaucoma.
   * Prove that the test product is as safe as the reference product in patients with primary open-angle glaucoma.

   Study design:

   A multicenter, prospective, open-label, randomized, comparative, controlled, parallel-arm study evaluating the efficacy and safety in patients with a specific disease.

   Study subjects: 118 patients (59 subjects in each group) with elevated intraocular pressure induced by primary open-angle glaucoma (POAG), males and females in the age bracket of 18 to 75 years conforming to the inclusion and exclusion criteria.

   Patients randomized: 118 Dropouts: 1 Per protocol population: 117 Safety population: 118

   Inclusion criteria:
   * Females or males in the age bracket of 18 to 75 years.
   * Established stage I and II primary open-angle glaucoma in one or both eyes.
   * IOP = 21-27 mm Hg (by Goldmann applanation tonometry).
   * Visual acuity 0.3 or better on the tested eye.
   * Patients who have signed an informed consent to participate in the study.
   * For females of child-bearing potential - a negative pregnancy test and consent to use reliable contraception methods throughout the study.

   Exclusion criteria:
   * Contraindications or hypersensitivity to the active ingredient (dorzolamide) or excipients.
   * The only eye.
   * Visual acuity ˂ 0.3 after correction.
   * An active infectious inflammatory process on the tested eye within 3 months prior to pre-study medical examination.
   * Pronounced visual field defects (III and IV stage open-angle glaucoma).
   * IOP ˃ 27 mm Hg or ˂ 21 mm Hg as at the IOP measuring at 10.00 a.m. (±1 h) in any of the eyes on the screening visit day.
   * Closed or nearly closed anterior chamber angle (ACA) or history of acute angle close.
   * Surgical and laser eye interventions over the last 3 months.
   * Manifest ocular media opacification hindering the treatment efficacy evaluation.
   * Other eye diseases that may affect dynamics of the parameters used for the treatment efficacy evaluation.
   * Inflammatory conditions of the eye and appendages (blepharitis, conjunctivitis).
   * Chronic kidney disease (creatinine clearance ˂ 30 mL/min).
   * Hyperchloremic acidosis.
   * Concomitant administration of oral carbonic anhydrase inhibitors.
   * Children and adolescents under 18 years.
   * The patient's participation in another clinical trial for the last 3 months.
   * Any systemic or mental disorder/condition (unmanageable arterial hypertension, decompensated diabetes mellitus, severe renal impairment) or clinically relevant abnormal laboratory tests at screening that, in the Investigator's opinion, may put a patient to a significant risk, or compromise the study results, or appreciably affect the possibility for the patient to participate in the study.
   * A patient who is unlikely to comply with the protocol requirements, e.g., is undisposed to cooperation, and is unlikely to complete the study.
   * Females and males of reproductive age refusing to use efficacious contraception methods.
   * Females during pregnancy and breastfeeding. Drug therapy type

   Test product:

   Trade name: Dorzol Active ingredient: dorzolamide Pharmaceutical form: eye drops Dosage: 20 mg/mL Posology and method of administration: Instillation into the conjunctival sac of 1 drop 3 times daily for 12 weeks.

   Manufacturer: JADRAN - GALENSKI LABORATORIJ d.d., Croatia

   Reference product description and labeling:

   Trade name: Trusopt® Active ingredient: dorzolamide Pharmaceutical form: eye drops Dosage: 20 mg/mL Posology and method of administration: 3 times daily Manufacturer: Laboratoires Merck Sharp & Dohme-Chibret, France Study duration: Screening: 7 days. The comparison product treatment lasted for 12 weeks (84±2 days). Follow-up period: 7 days. The overall study duration per patient did not exceed 99±2 days.

   The efficacy is established based on analysis of the parameters as follows:

   Primary endpoint

   • Mean IOP change from baseline.

   Secondary endpoints
   * IOP reduction rate to the target level of ≤ 18 mm Hg.
   * IOP reduction rate greater than 20%.
   * IOP reduction rate greater than 30%. Safety evaluation
   * Incidence of adverse events to a greater or lesser extent linked to the test or reference product, including those evaluated from laboratory test findings.
   * Treatment safety is evaluated from recording adverse events via analysis of complaints and symptoms, evaluation and interpretation of the findings of instrumental monitoring (biomicroscopy, ophthalmoscopy, IOP measures, perimetry) and laboratory tests.

   Statistical analysis Statistical analysis was performed using Statsoft Statistica Professional 13 and Microsoft Excel 2016 software.

   The Shapiro-Wilk test was used to evaluate the normality of distribution of quantitative attributes. Parametric tests were used for testing statistical hypotheses for parameters with the normal distribution, whereas nonparametric tests were used for parameters with the variance of the distribution. Student's t-test and Mann-Whitney U test were used for comparing the study groups in terms of quantitative attributes. The comparison of intragroup parameters before and after treatment was performed using the dependent samples t-test or the Wilcoxon test. The intragroup comparisons were also performed using nonparametric repeated measures ANOVA (the Friedman test). Qualitative attributes were analyzed using Pearson's χ2 test or Fisher's exact test (if the attribute incidence rate in at least one subgroup was ≤ 5).

   Statistically significant are differences with p-values < 0.05. Efficacy analysis of the comparison products provides for a conclusion on
   * Noninferiority of the test product Dorzol, eye drops (JADRAN - GALENSKI LABORATORIJ d.d., Croatia) vs. reference product Trusopt®, eye drops (Laboratoires Merck Sharp & Dohme-Chibret, France) by the primary endpoint:

     * No statistically significant intergroup differences have been observed regarding a mean intraocular pressure change from baseline either in the treatment or control group (p = 0.1609; Mann-Whitney U test).
     * The efficacy differences between the test and reference product by the primary criterion do not exceed the noninferiority margin of 1.5 mm Hg.

   Intergroup efficacy comparisons of the comparison products by the secondary endpoints have also been performed, with statistical significance of intergroup differences evaluated for ITT and PP populations:
   * ITT

     o No statistically significant intergroup differences have been observed regarding the IOP reduction rate to the target level of ≤ 18 mm Hg either in the treatment or control group (p = 0.5727; Pearson's χ2 test), which is indicative of Dorzol noninferiority by this parameter vs. reference product.

     o No statistically significant intergroup differences have been observed regarding the IOP reduction rate greater than 20% at visit 5 from baseline at visit 1 pre-dose either in the treatment or control group (p = 0.5661; Pearson's χ2 test), which is indicative of Dorzol noninferiority by this parameter vs. reference product.

     o No statistically significant intergroup differences have been observed regarding the IOP reduction rate greater than 30% at visit 5 from baseline at visit 1 pre-dose either in the treatment or control group (p = 0.4524; Pearson's χ2 test), which is indicative of Dorzol noninferiority by this parameter vs. reference product.
   * PP o No statistically significant intergroup differences have been observed regarding the IOP reduction rate to the target level of ≤ 18 mm Hg either in the treatment or control group (p = 0.5212; Pearson's χ2 test), which is indicative of Dorzol noninferiority by this parameter vs. reference product.

     o No statistically significant intergroup differences have been observed regarding the IOP reduction rate greater than 20% at visit 5 from baseline at visit 1 pre-dose either in the treatment or control group (p = 0.6494; Pearson's χ2 test), which is indicative of Dorzol noninferiority by this parameter vs. reference product.
     * No statistically significant intergroup differences have been observed regarding the IOP reduction rate greater than 30% at visit 5 from baseline at visit 1 pre-dose either in the treatment or control group (p = 0.4769; Pearson's χ2 test), which is indicative of Dorzol noninferiority by this parameter vs. reference product.

   The safety evaluation provided for the conclusions as follows:
   * Analysis of these AEs is indicative of comparable safety of the test product:

     o AE occurrence in the treatment group does not differ reliably from AE occurrence in the control group (p = 0.7058; Pearson's χ2 test).

     o AE link to the test product was most characterized as 'probable'; there were no statistically significant intergroup differences by this parameter either (p = 0,073).
     * AE severity was most characterized as mild; there were no statistically significant intergroup differences by this parameter either (p = 0.0863).
   * Analysis of the patients' laboratory test findings has identified statistically reliable differences by certain parameters (hemoglobin, ESR, AST, ALT, urea, total bilirubin, total protein, urine specific gravity). However, these differences are linked to patients' personality traits.

   Thus, based on all criteria specified in the Clinical Trial Protocol, the test product Dorzol and reference product Trusopt® demonstrate close efficacy and safety parameters. There are no statistically significant intergroup differences by any efficacy criteria tested. The efficacy differences between the test and reference product by the primary criterion do not exceed the noninferiority margin of 1.5 mm Hg. The above-stated provides for a conclusion on the test product Dorzol noninferiority vs. reference product Trusopt®.

ELIGIBILITY:
Inclusion Criteria:

* Females or males in the age bracket of 18 to 75 years.
* Established stage I and II primary open-angle glaucoma in one or both eyes.
* IOP = 21-27 mm Hg (by Goldmann applanation tonometry).
* Visual acuity 0.3 or better on the tested eye.
* Patients who have signed an informed consent to participate in the study.
* For females of child-bearing potential - a negative pregnancy test and consent to use reliable contraception methods throughout the study.

Exclusion Criteria:

* Contraindications or hypersensitivity to the active ingredient (dorzolamide) or excipients.
* The only eye.
* Visual acuity ˂ 0.3 after correction.
* An active infectious inflammatory process on the tested eye within 3 months prior to pre-study medical examination.
* Pronounced visual field defects (III and IV stage open-angle glaucoma).
* IOP ˃ 27 mm Hg or ˂ 21 mm Hg as at the IOP measuring at 10.00 a.m. (±1 h) in any of the eyes on the screening visit day.
* Closed or nearly closed anterior chamber angle (ACA) or history of acute angle close.
* Surgical and laser eye interventions over the last 3 months.
* Manifest ocular media opacification hindering the treatment efficacy evaluation.
* Other eye diseases that may affect dynamics of the parameters used for the treatment efficacy evaluation.
* Inflammatory conditions of the eye and appendages (blepharitis, conjunctivitis).
* Chronic kidney disease (creatinine clearance ˂ 30 mL/min).
* Hyperchloremic acidosis.
* Concomitant administration of oral carbonic anhydrase inhibitors.
* Children and adolescents under 18 years.
* The patient's participation in another clinical trial for the last 3 months.
* Any systemic or mental disorder/condition (unmanageable arterial hypertension, decompensated diabetes mellitus, severe renal impairment) or clinically relevant abnormal laboratory tests at screening that, in the Investigator's opinion, may put a patient to a significant risk, or compromise the study results, or appreciably affect the possibility for the patient to participate in the study.
* A patient who is unlikely to comply with the protocol requirements, e.g., is undisposed to cooperation, and is unlikely to complete the study.
* Females and males of reproductive age refusing to use efficacious contraception methods.
* Females during pregnancy and breastfeeding.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 118 (Actual)
Dates: Start 2017-04-05 (Actual); Primary Completion 2017-04-05 (Actual); Study Completion 2018-09-01 (Actual)

PRIMARY OUTCOMES:
Mean IOP change from baseline | 12 weeks
  Mean change in intraocular pressure (IOP) at visit 5 compared to baseline at visit 0

SECONDARY OUTCOMES:
IOP reduction rate to the target level of ≤ 18 mm Hg | 12 weeks
  Incidence of IOP reduction rate to the target level of ≤ 18 mm Hg (at visit 5)
IOP reduction rate by more than 20% | 12 weeks
  Incidence of IOP reduction rate by more than 20% (at visit 5)
IOP reduction rate by more than 30% | 12 weeks
  Incidence of IOP reduction rate by more than 30% (at visit 5)

CONTACTS AND LOCATIONS:
Overall Officials: Elmira Abdulaeva, PhD, Principal Investigator — Republican Clinical Ophthalmological Hospital of the Ministry of Health of the Republic of Tatarstan
Locations (1):
- State autonomous healthcare institution 'Republican Clinical Ophthalmological Hospital of the Ministry of Health of the Republic of Tatarstan', Kazan', Russia

IPD SHARING:
Plan to Share IPD: No